CLINICAL TRIAL: NCT06447844
Title: OsteoGen® Plug vs Freeze-dried Bone Allograft With Collagen Barrier for Alveolar Ridge Preservation (ARP): A Randomized Controlled Trial
Brief Title: OsteoGen Plug vs. Freeze-dried Bone Allograft With Collagen Barrier
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGuire Institute (Industry)
Collaborators: Impladent LTD (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OGP2024-01
Record Dates: First submitted 2024-05-29; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Nonterminal Premolar Needing Extraction

STUDY DESIGN:
Intervention Model Description: a multi-site, randomized, two-arm, controlled clinical trial using OsteoGen® Plug (Test) vs Freeze-dried Bone Allograft with collagen barrier
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- OsteoGen Plug (Experimental): OsteoGen® Plug (OGP) is a combination of bovine achilles tendon collagen matrix sourced from Australia or New Zealand and bioactive resorbable calcium apatite crystals intended for ARP. It is provided to clinicians in 3 different sizes to be placed in extraction socket.
  Interventions: Device: OsteoGen Plug
- BioGide (Active Comparator): This product is SOC treatment and will be used per packaging instructions.
  Interventions: Device: BioGide

INTERVENTIONS:
Device: OsteoGen Plug — OsteoGen® Plug is contoured to fill the three roots of the socket. Plug is delivered dry into a thoroughly debrided and actively bleeding socket. The OsteoGen® Plug is condensed firmly into the socket.
  Arms: OsteoGen Plug
Device: BioGide — BioGide is a resorbable collagen membrane
  Arms: BioGide

SUMMARY:
The study will be a multi-site, randomized, two-arm, controlled clinical trial using OsteoGen® Plug (Test) vs Freeze-dried Bone Allograft with collagen barrier (Control) for alveolar ridge preservation (ARP) in posterior extraction sites with intact buccal cortical plates.

DETAILED DESCRIPTION:
After tooth extraction and debridement, sockets will be packed with either test product (OGP), or control product (BioGide). Subjects will then undergo follow-up assessments conducted at day 7 (+3 days), day 14 (+3 days), and day 30 (+3 days) for oral exam, PROs, AEs, and complication assessments. Subjects will undergo follow-up assessments conducted at day 60 (+3 days) and day 90 (+3 days), for oral exam, PROs, AEs, complication assessments, standardized PA radiographs. Subjects will undergo follow-up assessments conducted at day 120 (+3 days) for oral exam, PROs, AEs, complication assessments, standardized PA radiograph, intraoral scan, and CBCT.

OPTIONAL Subjects will undergo follow-up assessments conducted at day 135 (+14 days) for oral exam, AEs, complication assessments, histologic core procurement, additional grafting assessment, prosthetic driven implant placement assessment.

Subjects will undergo follow-up assessments conducted at day 143 (+5 days) for oral exam, AEs, end of study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 to 75-yrs of age.
* Subjects with a nonterminal premolar in need of extraction with intention to pursue implant replacement.
* Proposed treatment site must have intact buccal cortical plates > 1 mm in thickness (buccal bone dehiscence up to 25% root length is permissible). Apical lesions are acceptable which do not perforate the cortical plate).
* Proposed treatment site must have intact adjacent natural teeth. (no adjacent edentulous sites or implants).
* Subjects can provide self-care (oral hygiene) without disabilities requiring assistance with daily oral hygiene measures.
* Subjects will have read, understood, and signed an institutional review board (IRB) approved Informed Consent Form (ICF).
* Subjects must be able and willing to follow study procedures and instructions.

Exclusion Criteria:

* Subjects with reported allergy or hypersensitivity to any of the products to be used in the study.
* Subjects with untreated / active periodontal disease.
* Subjects with vesiculobullous processes or other similar chronic oral lesions / conditions resulting in gingival irritation, discomfort/pain, or erosions.
* Tobacco/Cannabis users including cigarettes, vape, cigars, or smokeless tobacco.
* Uncontrolled medical conditions (e.g., diabetes mellitus, hypertension, cancer)
* Subjects who are lactating or pregnant or planning to become pregnant through their projected study duration.
* Subjects who would require a tissue supported interim prosthesis i.e. acrylic / valplast RPD (tooth supported interim prostheses i.e. essix retainers are acceptable)
* Subjects with long-term history of oral bisphosphonates (> 10 years).
* Subjects with a history of intravenous bisphosphonates.
* Subjects taking medications known to affect gingival conditions. (e.g., hyperplasia)
* Subjects taking corticosteroids or immunosuppressants on a regular basis prior to baseline examination.
* Subjects taking anticoagulant medications such as warfarin or Plavix or Eliquis who are not medically cleared to hold medication prior to and during procedure.
* Subjects participating in other clinical studies involving therapeutic intervention (either medical or dental).
* Subjects, who in the opinion of the investigator, for any reason other than those listed above, will not be able to complete the study per protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-07-28 (Estimated); Study Completion 2029-11-28 (Estimated)

PRIMARY OUTCOMES:
New bone formation | 120 days
  new bone formation will be determined by Cone Beam Cat Scan (CBCT) at Day 120

SECONDARY OUTCOMES:
Change in ridge height compared to screening as determined by Cone Beam Cat Scan (CBCT) | 120 days
  two CBCTs will be compared, one from screening, the other at 120 days.

OTHER OUTCOMES:
Change in ridge width compared to screening at 3mm and 5mm below crest | 120 days
  two CBCTs will be compared, one from screening, the other at 120 days.
Volumetric analysis of soft tissue/ridge height and width via intraoral scans | 120 days
  Intraoral scans will be compared to baseline, pre-surgery and 120 days.
Histologic assessment of NBF (new bone formation), RG (residual graft particle) and connective tissue at 4 months if implant is placed | 4 months post implant placement
  histology samples will be collected 4 months post implant placement for analysis on bone growth,
wound closure assessment | 120 days
  wound closure will be assessed at all post surgical visits.
number of treatment sites requiring additional grafting at time of implant placement | During procedure (time of implant placement)
  oral exam of dentition to determine if any additional grafting is needed to treatment sites.
cost effectiveness analysis | 120 days
  comparison of experimental procedure vs. standard treatment.
baseline buccal plate thickness influence on outcomes | 120 days
  buccal plate thickness documented by CBCT will be compared to outcomes.
change in phenotype | 120 days
  the change in soft and hard tissue thickness supporting structures of the teeth.
time comparison between treatment groups from post extraction to ARP procedure completion (final suture) | surgical visit
  time will be document for both arms from start of surgery to last suture being placed
Change in ridge width compared to screening at crest as determined by CBCT. Change in ridge width compared to baseline screening at crest as determined by CBCT. Change in ridge width compared to screening at crest as determined by CBCT. | 120 days
  two CBCTs will be compared, one from screening, the other at 120 days.
complication type and incidence rates | 120 days
  complications will be collected at all visits post surgery
Prosthetic driven implant feasibility assessment | 120 days
  a determination if implant could have been placed without additional grafting.
Safety and tolerability/biocompatibility:Adverse events | 120 days
  adverse events will be collected from baseline visit through end of study
Patient demographics and robust health history influence outcomes | 120 days
  patient demographics will be collected at screening and compared to outcomes at Day 120
Patient reported outcomes (pain, satisfaction) | 120 days
  PROs will be collected from baseline to day 120 to determine level of pain on a scale from 1 (no discomfort) to 10 (as much discomfort as i have ever felt) and satisfaction on a scale of 0 (completely dissatisfied) to 10 (completely satisfied).
Clinician reported outcomes for usability (ease of use, time for each graft procedure, site vascularity) | visit 2 post surgery
  clinicians will be asked to provide their opinions on useability of each product. Ease of use scale 0 (completely dissatisfied) to 10 (completely satisfied) and vascularity rating from 1 (avascular blood flow) to 5 (blood flow readily apparent without cortical penetration)
Long term implant assessments | post implant placement (outside of study after 120 days)
  optional assessment if an implant is placed at some point in the future.Details not yet specified.
histology cores if implant placement in future | post implant placement (outside of study after 120 days)
  optional additional histology assessments may be done if implant is placed at some point in the future.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - McClain and Schallhorn Periodontics and Implant Dentistry, Aurora, Colorado
  - Colorado Gum Care, Broomfield, Colorado
  - The Perio Studio, Boston, Massachusetts
  - Seven Lakes Periodontics, Fenton, Michigan
  - Perio & Implant Associates of Middle TN, Nashville, Tennessee
  - Perio Health Professionals, Houston, Texas
  - Gulf Coast Periodontics, Victoria, Texas
  - WisNova Institute of Dental Specialists, Kenosha, Wisconsin